CLINICAL TRIAL: NCT04619303
Title: A Randomized Clinical Trial of Intravitreal dexamethasOne Versus Bevacizumab in Aboriginal and Torres Strait Islander patientS With Diabetic Macular Oedema (The OASIS Study)
Brief Title: Intravitreal Dexamethasone vs Bevacizumab in Aboriginal People With DMO
Acronym: OASIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lions Eye Institute, Perth, Western Australia (Other)
Collaborators: Lions Outback Vision (Unknown); Allergan (Industry)
Responsible Party: Principal Investigator, A/Prof. Hessom Razavi, Associate Professor, Lions Eye Institute, Perth, Western Australia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OASIS
Record Dates: First submitted 2020-10-27; First posted 2020-11-06 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
Keywords: Diabetic macular edema; Aboriginal; Australian
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Dexamethasone; Calcium Dobesilate; Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone Implant (Experimental): Receive 0.7mg dexamethasone implant (Ozurdex) at baseline visit. Monthly review with repeat administration of intravitreal treatment every three months for DMO and laser as clinically indicated.
  Interventions: Drug: Dexamethasone intravitreal implant
- Bevacizumab (Active Comparator): Receive 1.25mg/0.05ml bevacizumab (Avastin) at baseline visit. Monthly review with repeat administration of intravitreal treatment every one month for DMO and laser as clinically indicated.
  Interventions: Drug: Bevacizumab Injectable Product

INTERVENTIONS:
Drug: Dexamethasone intravitreal implant — Intravitreal injection of 0.7mg dexamethasone implant
  Other Names: Ozurdex; DEX-implant
  Arms: Dexamethasone Implant
Drug: Bevacizumab Injectable Product — Invtravitreal injection of 1.25mg/0.05mL bevacizumab
  Other Names: Avastin
  Arms: Bevacizumab

SUMMARY:
DMO is the most common cause of visual loss in people with diabetes. Regular injections of bevacizumab (Avastin) given as frequently as every month remain the current standard of care for centre-involving DMO; however, this regimen is impractical for many Aboriginal patients. Using Ozurdex implants every 3-6 months could be as effective as the currently used Avastin injections. In order to address this real-world problem, this study seeks to investigate whether it is possible to safely use a long-acting steroid preparation such as the dexamethasone IVT implant (Ozurdex) to manage DMO in Aboriginal patients living in Western Australia.

DETAILED DESCRIPTION:
The prevalence of self-reported DM in Aboriginal Australians is reported to be as high as 38%. Despite gradual improvements in underlying social determinants of health, the high morbidity and mortality attributed to DM in Aboriginal populations indicates significant ongoing issues with adherence to screening and treatment regimens. The greater prevalence of DM in the Aboriginal Australian population would be expected to account (at least in part) for the observed complication rates, including DR.

DMO is characterised by swelling of the central retina. The hypoxic retinal conditions in diabetic individuals result in structural changes in the vessel walls and a functional impairment of the blood-retinal barrier. The resultant increase in vascular permeability causes retinal oedema, and loss of central vision ensues when oedema involves the macula. Treatment is aimed at reducing visual loss by targeting factors involved in the activated hypoxia pathway, or with laser targeting dysfunctional blood vessels to limit leakage. Laser was the first treatment shown to effectively reduce DMO and improve vision; however, it cannot be applied to the very centre of the macula. More recently, DMO has been shown to respond to intraocular injections with anti-VEGF agents (bevacizumab, ranibizumab, and aflibercept), reducing reliance on laser treatments.

Corticosteroids are anti-inflammatory agents with anti-VEGF and anti-proliferative effects. Unfortunately, the increased rates of cataract and elevated IOP are the main adverse effects of the IVT corticosteroid treatments, including triamcinolone, making this a less-appealing option than anti-VEGF agents. However, their efficacy has been demonstrated in a subgroup of pseudophakic patients with DMO, where triamcinolone plus laser treatment was shown to be superior to laser treatment alone, and equivalent to ranibizumab (alone or with laser treatment). First-line treatment with triamcinolone is also the most cost-effective option for pseudophakic patients. Thus, IVT triamcinolone is considered one of the effective adjunct modalities for the treatment of DMO and has emerged as an alternative therapy to anti-VEGF agents for persistent or refractory DMO.

Ozurdex (Allergan, Irvine, CA, United States) is a unique biodegradable dexamethasone IVT implant. This slow-release preparation of dexamethasone (a highly potent steroid with a short half-life) has greater long-term efficacy than conventional forms of IVT triamcinolone, with the IVT concentration peaking within 3 months and sustained for up to 6 months post injection. This translates clinically to less frequent injections than conventional treatment with monthly IVT triamcinolone. The geography and population being studied in this trial create some unique challenges, which demand a more flexible study protocol. Longer-acting IVT agents such as Ozurdex have the potential to significantly improve DMO-associated visual morbidity with greater feasibility when used for Aboriginal patients with or at risk of DMO.

ELIGIBILITY:
Inclusion criteria:

* Self-identifying as Aboriginal Australian or Torres Strait Islander
* Adults aged 18 years and over
* Diagnosis of DM (type 1 or type 2)
* BCVA of at best 0.2 LogMAR (20/32) 6/9 in the study eye
* Pseudophakic, or phakic with significant lens opacity and scheduled to undergo cataract surgery at the time of enrolment
* Presence of any grade of DR with centre-involving DMO, as defined by clinical examination and OCT scan findings

  * Active DMO: Centre-involving/threatening DMO, as defined by clinical examination and OCT scan findings.
  * At risk of DMO: Patients scheduled for cataract surgery with non-centre involving DMO who are assessed as being at risk of post-operative centre-involving DMO based on clinical examination, OCT scan findings, and Investigator discretion.

Exclusion criteria:

* Intervention: Previous treatment in the study eye including at the time of the first trial treatment with:

  * IVT anti-VEGF injections within the last six weeks;
  * Macular laser treatment within the last four months;
  * IVT triamcinolone or triescence within the last six months; at the time of the first trial treatment.
* History of open-angle glaucoma or steroid-induced IOP elevation that required IOP-lowering treatment or, IOP ≥25 (Goldmann applanation) on two consecutive clinic visits.
* Eyes with concurrent ocular pathology other than DMO, or a cataract-causing visual loss, including macular ischaemia as determined by clinical examination and FFA imaging.
* Women who are breastfeeding, confirmed as pregnant or planning on becoming pregnant in the next 6-12 months.
* Participants for whom Ozurdex or Avastin treatment are contraindicated as per product information:

  * Active or suspected ocular/periocular infections, including most viral diseases of the cornea and conjunctiva, active epithelia herpes simplex keratitis (dendritic keratitis), vaccinia, varicella, mycobacterial infections, and fungal diseases.
  * Aphakic eyes with rupture of the posterior lens capsule.
  * Eyes with an anterior chamber intraocular lens and rupture of the posterior lens capsule.
  * Known angina, myocardial infarction, TIA or CVA in the last three months.
  * Known hypersensitivity to any components of these products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Difference in best corrected visual acuity change between treatment arms | 12 months
  The primary outcome measure will be the difference in the BCVA change from baseline to 12 months between treatment arms, with a non-inferiority margin of 0.1 LogMAR (equivalent to one line of Snellen visual acuity). The BCVA will be measured for all study participants at each clinic visit.

SECONDARY OUTCOMES:
Best corrected visual acuity loss or gain | 12 months
  The proportion of participants with a BCVA loss or gain of <0.3 LogMAR (termed 'stable BCVA'), a BCVA loss of ≥0.3 LogMAR ('decline in BCVA'), or a BCVA gain of ≥0.3 LogMAR ('gain in BCVA').
Change in central macular thickness | 12 months
  Change in the CMT from baseline to 12 months as measured by OCT.
Number of injections | 12 months
  Number of IVT injections given per participant.
Appointments attended | 12 months
  Number of appointments attended per participant.
Intraocular pressure change | 12 months
  The change in the mean IOP.
Intraocular pressure elevation | 12 months
  The number of participants with one or more occasions of IOP elevation >28 mmHg.
Intraocular pressure elevation requiring treatment | 12 months
  IOP elevation requiring medical, laser or surgical treatment.
Adverse Events | 12 months
  Adverse events (AEs), serious adverse events (SAEs) and serious adverse reactions (SARs) coded according to the National Medical Research Council (2016) safety monitoring and reporting in clinical trials definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Angus Turner, FRANZCO, Study Director — Lions Eye Institute
Locations (13):
- Australia (13):
  - Broome Regional Aboriginal Medical Service, Broome, Western Australia
  - Derby Hospital, Derby, Western Australia
  - Fitzroy Crossing Hospital, Fitzroy Crossing, Western Australia
  - Halls Creek Health Service, Halls Creek, Western Australia
  - Bega Garnbirringu Health Service, Kalgoorlie-Boulder, Western Australia
  - Nickol Bay Hospital, Karratha, Western Australia
  - Ord Valley Aboriginal Health Service, Kununurra, Western Australia
  - Laverton Hospital, Laverton, Western Australia
  - Derbarl Yerrigan Health Service Inc., Perth, Western Australia
  - Lions Eye Institute Nedlands, Perth, Western Australia
  - Lions Eye Institute Midland, Perth, Western Australia
  - Mawarnkarra Health Service, Roebourne, Western Australia
  - Wirraka Maya Health Service Aboriginal Corporation, South Hedland, Western Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data as well as visit data with primary and secondary outcome data and accompanying data dictionary will be made available.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 6 months

REFERENCES:
- [Background] Xie J, Arnold AL, Keeffe J, Goujon N, Dunn RA, Fox S, Taylor HR. Prevalence of self-reported diabetes and diabetic retinopathy in indigenous Australians: the National Indigenous Eye Health Survey. Clin Exp Ophthalmol. 2011 Aug;39(6):487-93. doi: 10.1111/j.1442-9071.2011.02502.x. Epub 2011 Mar 24. PMID 21819502
- [Background] Kaidonis G, Mills RA, Landers J, Lake SR, Burdon KP, Craig JE. Review of the prevalence of diabetic retinopathy in Indigenous Australians. Clin Exp Ophthalmol. 2014 Dec;42(9):875-82. doi: 10.1111/ceo.12338. Epub 2014 May 5. PMID 24666566
- [Background] Wong J, Molyneaux L, Constantino M, Twigg SM, Yue DK. Timing is everything: age of onset influences long-term retinopathy risk in type 2 diabetes, independent of traditional risk factors. Diabetes Care. 2008 Oct;31(10):1985-90. doi: 10.2337/dc08-0580. Epub 2008 Jul 15. PMID 18628565
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Progression of retinopathy with intensive versus conventional treatment in the Diabetes Control and Complications Trial. Diabetes Control and Complications Trial Research Group. Ophthalmology. 1995 Apr;102(4):647-61. doi: 10.1016/s0161-6420(95)30973-6. PMID 7724182
- [Background] Wong TY, Mwamburi M, Klein R, Larsen M, Flynn H, Hernandez-Medina M, Ranganathan G, Wirostko B, Pleil A, Mitchell P. Rates of progression in diabetic retinopathy during different time periods: a systematic review and meta-analysis. Diabetes Care. 2009 Dec;32(12):2307-13. doi: 10.2337/dc09-0615. PMID 19940227
- [Background] Klein R, Klein BE. Blood pressure control and diabetic retinopathy. Br J Ophthalmol. 2002 Apr;86(4):365-7. doi: 10.1136/bjo.86.4.365. No abstract available. PMID 11914198
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Michaelides M, Kaines A, Hamilton RD, Fraser-Bell S, Rajendram R, Quhill F, Boos CJ, Xing W, Egan C, Peto T, Bunce C, Leslie RD, Hykin PG. A prospective randomized trial of intravitreal bevacizumab or laser therapy in the management of diabetic macular edema (BOLT study) 12-month data: report 2. Ophthalmology. 2010 Jun;117(6):1078-1086.e2. doi: 10.1016/j.ophtha.2010.03.045. Epub 2010 Apr 22. PMID 20416952
- [Background] Diabetic Retinopathy Clinical Research Network; Elman MJ, Aiello LP, Beck RW, Bressler NM, Bressler SB, Edwards AR, Ferris FL 3rd, Friedman SM, Glassman AR, Miller KM, Scott IU, Stockdale CR, Sun JK. Randomized trial evaluating ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2010 Jun;117(6):1064-1077.e35. doi: 10.1016/j.ophtha.2010.02.031. Epub 2010 Apr 28. PMID 20427088
- [Background] Elman MJ, Bressler NM, Qin H, Beck RW, Ferris FL 3rd, Friedman SM, Glassman AR, Scott IU, Stockdale CR, Sun JK; Diabetic Retinopathy Clinical Research Network. Expanded 2-year follow-up of ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2011 Apr;118(4):609-14. doi: 10.1016/j.ophtha.2010.12.033. PMID 21459214
- [Background] Dewan V, Lambert D, Edler J, Kymes S, Apte RS. Cost-effectiveness analysis of ranibizumab plus prompt or deferred laser or triamcinolone plus prompt laser for diabetic macular edema. Ophthalmology. 2012 Aug;119(8):1679-84. doi: 10.1016/j.ophtha.2012.01.049. Epub 2012 Apr 13. PMID 22503301
- [Background] Al Dhibi HA, Arevalo JF. Clinical trials on corticosteroids for diabetic macular edema. World J Diabetes. 2013 Dec 15;4(6):295-302. doi: 10.4239/wjd.v4.i6.295. PMID 24379920
- [Background] Chew EY, Benson WE, Remaley NA, Lindley AA, Burton TC, Csaky K, Williams GA, Ferris FL 3rd. Results after lens extraction in patients with diabetic retinopathy: early treatment diabetic retinopathy study report number 25. Arch Ophthalmol. 1999 Dec;117(12):1600-6. doi: 10.1001/archopht.117.12.1600. PMID 10604663
- [Background] Cetin EN, Yildirim C. Adjuvant treatment modalities to control macular edema in diabetic patients undergoing cataract surgery. Int Ophthalmol. 2013 Oct;33(5):605-10. doi: 10.1007/s10792-012-9695-1. Epub 2012 Dec 18. PMID 23248073
- [Background] Chang-Lin JE, Attar M, Acheampong AA, Robinson MR, Whitcup SM, Kuppermann BD, Welty D. Pharmacokinetics and pharmacodynamics of a sustained-release dexamethasone intravitreal implant. Invest Ophthalmol Vis Sci. 2011 Jan 5;52(1):80-6. doi: 10.1167/iovs.10-5285. PMID 20702826
- [Background] Zalewski D, Raczynska D, Raczynska K. Five-month observation of persistent diabetic macular edema after intravitreal injection of Ozurdex implant. Mediators Inflamm. 2014;2014:364143. doi: 10.1155/2014/364143. Epub 2014 Feb 10. PMID 24659860
- [Background] Dutra Medeiros M, Postorino M, Navarro R, Garcia-Arumi J, Mateo C, Corcostegui B. Dexamethasone intravitreal implant for treatment of patients with persistent diabetic macular edema. Ophthalmologica. 2014;231(3):141-6. doi: 10.1159/000356413. Epub 2013 Dec 19. PMID 24356099
- [Background] Zucchiatti I, Lattanzio R, Querques G, Querques L, Del Turco C, Cascavilla ML, Bandello F. Intravitreal dexamethasone implant in patients with persistent diabetic macular edema. Ophthalmologica. 2012;228(2):117-22. doi: 10.1159/000336225. Epub 2012 Feb 3. PMID 22310491
- [Background] Haller JA, Kuppermann BD, Blumenkranz MS, Williams GA, Weinberg DV, Chou C, Whitcup SM; Dexamethasone DDS Phase II Study Group. Randomized controlled trial of an intravitreous dexamethasone drug delivery system in patients with diabetic macular edema. Arch Ophthalmol. 2010 Mar;128(3):289-96. doi: 10.1001/archophthalmol.2010.21. PMID 20212197
- [Background] Boyer DS, Faber D, Gupta S, Patel SS, Tabandeh H, Li XY, Liu CC, Lou J, Whitcup SM; Ozurdex CHAMPLAIN Study Group. Dexamethasone intravitreal implant for treatment of diabetic macular edema in vitrectomized patients. Retina. 2011 May;31(5):915-23. doi: 10.1097/IAE.0b013e318206d18c. PMID 21487341
- [Background] Hariprasad SM, Mieler WF, Grassi M, Green JL, Jager RD, Miller L. Vision-related quality of life in patients with diabetic macular oedema. Br J Ophthalmol. 2008 Jan;92(1):89-92. doi: 10.1136/bjo.2007.122416. Epub 2007 Jun 21. PMID 17584999
- [Background] Chen E, Looman M, Laouri M, Gallagher M, Van Nuys K, Lakdawalla D, Fortuny J. Burden of illness of diabetic macular edema: literature review. Curr Med Res Opin. 2010 Jul;26(7):1587-97. doi: 10.1185/03007995.2010.482503. PMID 20429823
- See also: Australian Bureau of Statistics. Diabetes in Australia: A Snapshot, 2007-08. Cat. no. 4820.0. — https://www.abs.gov.au/ausstats/abs@.nsf/Lookup/4820.0.55.001Media+Release12007-08

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/03/NCT04619303/Prot_SAP_000.pdf